CLINICAL TRIAL: NCT02653222
Title: Feasibility Study of Perivascular Computer Tomography-guided Ethanol Sympatholysis for the Treatment of Therapy-resistant Arterial Hypertension
Brief Title: Chemical Renal Ethanol Sympatholysis Under CT Guidance Use for the Control of Therapy-Resistant Hypertension
Acronym: SCRATCH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: patient recruitment is difficult
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC15.182; 2015-002579-59 (EudraCT Number)
Record Dates: First submitted 2016-01-05; First posted 2016-01-12 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Hypertension Resistant to Conventional Therapy; Kidney Failure, Chronic
Keywords: Ethanol Sympathicolysis; Computer Tomography guidance; Denervation; Kidney Transplantation; Dialysis
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Kidney Failure, Chronic | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal sympathicolysis (Experimental): The patient will have:
  1. Ambulatory Blood Pressure Monitoring
  2. Magnetic Resonance Angiography
  3. Blood test
  4. Renal sympathicolysis
  5. Ambulatory Blood Pressure Monitoring
  6. Magnetic Resonance Angiography
  Interventions: Procedure: Renal sympathicolysis; Procedure: Ambulatory Blood Pressure Monitoring; Radiation: Magnetic Resonance Angiography; Biological: Blood test

INTERVENTIONS:
Procedure: Renal sympathicolysis
  Other Names: renal sympathetic denervation; CT guidance
Procedure: Ambulatory Blood Pressure Monitoring — 1 month before and after surgery the patient will have an ABPM over 24h
  Other Names: ABPM
Radiation: Magnetic Resonance Angiography — 1 month before and after surgery the patient will have a MRA
  Other Names: MRA
Biological: Blood test — complete blood count, blood platelets, coagulation profile, irregular agglutinins search

SUMMARY:
In this study the investigators are going to assess the feasibility of this innovate technique of renal sympathetic denervation by translumbar access under ct-guidance.

To limit the potential impact on the kidney, the investigators chose a population of chronic renal failure patients on dialysis or renal transplant (with native kidneys still present) and having resistant treatment hypertension despite antihypertensive combination therapy well conducted.

The investigators expect to obtain a decrease of the blood pressure at the 24-hours ambulatory blood pressure monitoring (ABPM) one month after the sympathetic denervation.

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old,
* patient with triple antihypertensive therapy (maximum tolerated dose) with a diuretic, except for anuric patients, and without modification treatment:
* in the last two months,
* expected in the next three months,
* renal transplanted patients with native kidneys followed for hypertension before transplant, and having a arterial systolic pressure ≥ 160 mmHg on the average of 3 measurements taken during the screening consultation and during at least one previous consultation OR
* chronic renal failure patient with dialysis and having a arterial systolic pressure ≥ 160 mmHg on the average of 3 measurements taken during the screening consultation and during at least one previous consultation
* patient affiliated to social security or similarly regime
* patient who signed the consent to participate in the study

No Inclusion Criteria:

* renal artery anatomy against-indicating the procedure including:
* 3 homolateral renal arteries
* kidney surgery including bypass surgery or renal artery reimplantation
* volume-dependent type of hypertension
* secondary hypertension (not included nephropathy)
* orthostatic hypotension associated with symptoms during the previous year
* medical history including:

  * acute coronary syndrome, unstable angina, stroke within 6 months preceding the period of inclusion,
  * surgery scheduled on the kidney, the renal arteries or the retroperitoneum during patient participation in the study period
  * chronic alcoholism
* anticoagulants or antiplatelet agents for which a therapeutic window can not be considered (except aspirin dose less than or equal to 160mg / day)
* contraindication to the realization of an MRI
* included in another trial assessing a medicament or a medical device or a surgical procedure
* protected person referred to in Articles L1121-5 to L1121-8 of the Code of Public Health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Success or failure of the peri-arterial technique injection of ethanol under CT guidance. | 2 hours
  Assess the technical feasibility of a new procedure of renal denervation chemical sympatholysis with ethanol, by a translumbar access, guided by CT, in a population of chronic dialysis or transplant failure patients followed for resistant treatment hypertension.
  The measure is a score based on the distribution of the ethanol near the aorta-renal angle

SECONDARY OUTCOMES:
Any clinical adverse event, radiological or biological related to the procedure and between it and the end of the study (MRI and follow up to 1 month). | One month
  Assess the occurrence of adverse events in the population who received the intervention by chemical sympatholysis during the month following the intervention
Change of the blood pressure between baseline and 1 month after surgery The results of this difference is in mmHg. | baseline at one month before surgery and 1 month after surgery
  Assess the effect of the chemical kidney sympatholysis on blood pressure one month after surgery.
Duration of the procedure between the first scanner acquisition and the latest acquisition of control. The result is in minutes. | 2 hours
  Assess the duration of the chemical sympatholysis procedure by translumbar access under CT guidance
A score will be established with one point by angle aorto-renal upper cover and one point on each quarter of the circumference of renal artery covered with ethanol. | One month
  Assess at 1 month follow up the chemical sympatholysis effect on blood pressure based on the distribution of ethanol (visualized by prior injection of contrast medium).

CONTACTS AND LOCATIONS:
Overall Officials: Julien Ghelfi, Md, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - University Hospital, Grenoble, Isère
  - Grenoble Association for the Dialysis of Uremic Chronicles, La Tronche, Isère

IPD SHARING:
Plan to Share IPD: No